CLINICAL TRIAL: NCT05210738
Title: A Cohort Observational Study Comparing the Outcomes of Single-incision Sling vs Urethral Bulking During Prolapse Surgery for Occult Stress Incontinence
Brief Title: Single-incision Sling vs Urethral Bulking During Prolapse Surgery for Occult Stress Incontinence
Status: Completed | Type: Observational
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Abdelaziz, MD, The Christ Hospital
Other Study IDs: E21-53
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Single incision sling group: The patient will receive Altis mini-incision sling for treatment of occult SUI
  Interventions: Device: Single incision sling
- Urethral bulking group: The patient will receive Bulkamid urethral bulking agent for treatment of SUI
  Interventions: Drug: Bulkamid bulking agent

INTERVENTIONS:
Device: Single incision sling — Single incision sling is used to treat occult SUI
  Groups: Single incision sling group
Drug: Bulkamid bulking agent — Urethral bulking by Bulkamid is used to treat occult SUI
  Groups: Urethral bulking group

SUMMARY:
The aim is to compare outcomes of two different procedures to prevent occult stress urinary incontinence (SUI) in patients who are having pelvic organ prolapse surgeries

DETAILED DESCRIPTION:
The aim is to compare outcomes of two different procedures to prevent occult stress urinary incontinence (SUI) in patients who are having pelvic organ prolapse surgeries. Charts will be reviewed for patients who had single- incision sling or urethral bulking injection with other prolapse surgeries to address occult stress incontinence at The Christ Hospital from the period of January 2019 to June 2021. Patients who didn't have any occult stress incontinence pre-operatively and didn't receive any anti-incontinence procedure during their prolapse surgery will be included as a control group. Surgical details, adverse events and postoperative voiding times will be collected from the chart. Patients will be contacted by a telephone to administer a validated questionnaire; a 3-day bladder diary to quantify urinary incontinence will be send to the patient to complete and return by mail.

The purpose of the study is to investigate whether urethral bulking is as effective as single- incision sling in treating occult stress incontinence.

ELIGIBILITY:
Inclusion Criteria:

* -Females who are 18 years or old who were scheduled to either urethral bulking (Bulkamid) or single-incision sling (Altis sling) to address occult SUI with prolapse surgery. All patients reported no history of SUI preoperatively and during office physical exam, positive SUI was demonstrated during prolapse reduction.
* Females who are 18 years or old who didn't have occult stress incontinence before their prolapse surgery and didn't receive any stress incontinence surgery during their prolapse surgery during the same period will be included as a control group.
* English speaking patients.

Exclusion Criteria:

* Patients who had either single-incision sling or urethral bulking with documented preoperative history of stress incontinence. Patients with a history of previous surgery for SUI.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced prolapse and preoperative evaluation showed occult stress incontinence
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Urinary Distress Inventory, Short Form (UDI-6) | one year after surgery
Incontinence Impact Questionnaire, Short Form (IIQ-7) | one year after surgery
Voiding diary | one year after surgery

SECONDARY OUTCOMES:
The rate of complications in both groups which includes adverse events, rate of urine retention with prolonged catheterization, and UTI. | one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelaziz, Principal Investigator — The Christ Hospital
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No